CLINICAL TRIAL: NCT03532269
Title: Validation of the Sleep Assessment Algorithm in the Medical Application Nightly and Comparing it to Polysomnography in 24 Healthy Individuals
Brief Title: Validation of the Sleep Assessment Algorithm in the Medical Application Nightly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamJay Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 001_Nightly_2017
Record Dates: First submitted 2017-10-16; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Sleep Disorder; Nightmare
Keywords: sleep; nightmare; app
MeSH Terms: conditions — Sleep Wake Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: 3rd night with acoustic stimulation (Experimental): Arm A: PSG (3 nights) with Nightly App - acoustic stimulation during the 3rd night.
  Interventions: Device: Nightly App
- B: 2nd night with acoustic stimulation (Experimental): Arm B: PSG (3 nights) with Nightly App - acoustic stimulation during the 2nd night.
  Interventions: Device: Nightly App

INTERVENTIONS:
Device: Nightly App — The Nightly application will be installed independently on the user's smartphone. Once the user has set up their account and has logged in, they can then perform regular sleep quality assessments. In order to record a measurement, the user must first select a film (first screen) and watch it (second screen), the visualizations and acoustics aid in the process of falling asleep. After the film finishes, the participant places the phone on the corner of the bed, firstly with the screen facing up, and then under his/her pillow. Throughout the night, the application registers sleep phases that will be analyzed later.

SUMMARY:
The Nightly medical application prototype is a potential, non-invasive class I medical device. The application has the potential to combine both diagnostic and therapeutic procedures for sleep. At home, Nightly measures the user's motion during sleep and then records the sleep pattern from the received data. The obtained data are then used for the diagnosis of sleep disorders (REM and NREM sleep). Using acoustic and visual stimulation, the application has the capability to support the natural process of falling asleep, provide a better night's sleep by minimizing sleep deprivation and nightmares, while awakening the user at the appropriate moment (during light sleep).

DETAILED DESCRIPTION:
The study is a cohort, single-center, randomized trial. The duration of one participant included in the study is three successive nights. Visual analysis of polysomnographic recordings taken from the second and third nights will be performed independently by two independent, blinded experts. According to the sleep architecture description derived from the Nightly application, polysomnographic and actigraphy studies will be assessed using the intraclass correlation coefficient, ICC, version "Two-Way Random". Parameters of the sleep architecture will be the average total length of the individual sleep phases (provided with standard deviations and coefficients of variability defined as the quotient of standard deviation and mean).

ELIGIBILITY:
Inclusion Criteria:

Any healthy individual who meets all the following criteria may be included in the study:

1. Age 18 to 40 years.
2. Signed Informed Consent Form for participation in the study
3. No chronic illnesses (A medical interview will be conducted during the participants first visit)
4. Does not take any medication chronically (According to the medical interview with the participants during the first visit)

Exclusion Criteria:

A person who meets any one of the following criteria cannot be included in the study:

1. Primary sleep disorders. (An in-depth medical interview during the first visit to be supplemented with: Holland Sleep Disorders Questionnaire which evaluates the risk of primary sleep disorders according to the International Classification of Sleep Disorders (ICSD-3), Athens insomnia scale which assesses the risk of insomnia and the STOP-BANG scale, evaluates the risk for sleep apnea; a journal will also be kept noting dreams between the first and second visit.
2. History of cancer or active cancer.
3. Disorders of the nervous system (e.g. epilepsy, migraine).
4. Mental disorders (e.g. depression, bipolar disorder, schizophrenia).
5. Active infection during the study. (Medical history, body temperature measurement and physical examination)
6. Consuming within 12 hours preceding the sleep examination: coffee, caffeinated teas or other beverages containing caffeine, caffeine, or other stimulants.
7. Consuming alcohol on the day of the examination.
8. Pregnancy and lactation (based on the patient's own declaration, pregnancy test is not planned prior to the examination).
9. Any contraindications to participate in the examination in the Investigator's opinion.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 15 M, 15 F
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
The ICC for distribution of the total duration of standby periods during phases NREM and REM | Through study completion - after 3rd night of PSG
  The ICC for distribution of the total duration of standby periods during phases NREM and REM should not be less than 0.6 in the comparative analysis of results provided by the Nightly application and at least one of the visual recordings from polysomnography.

SECONDARY OUTCOMES:
The ICC value when evaluating the accuracy of recognizing sleep phases and vigilance using the Nightly application | Through study completion - after 3rd night of PSG
  The ICC value when evaluating the accuracy of recognizing sleep phases and vigilance using the Nightly application and the reference method should be no less than the ICC when comparing actigraphy and the reference method
The incidence of arousal and wakening's | Through study completion - after 3rd night of PSG
  The stimulation produced by the Nightly application should not significantly affect the incidence of arousal and wakening's (when compared to analogous conditions without stimulation) with presumed statistical significance (p = 0.05). In other words, the aim of the experiment is to provide evidence that the distribution of arousals and wakening's measured in the study without stimulation is not statistically different from the distribution of the number of events during the Nightly application stimulation session
Evaluate the effect of acoustic stimulation - total sleep time | Through study completion - after 3rd night of PSG
  Total sleep time will be measured.
Evaluate the effect of acoustic stimulation - wake after sleep onset | Through study completion - after 3rd night of PSG
  Wake after sleep onset will be measured.
Evaluate the effect of acoustic stimulation - sleep latency | Through study completion - after 3rd night of PSG
  Sleep latency will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Jernajczyk, PhD, Principal Investigator — Institute of Neurology and Psychiatry
Locations (1):
- Institute of Psychiatry and Neurology in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No